CLINICAL TRIAL: NCT03276325
Title: Epidural Steroids Combined With Intrathecal Nalbuphine: Analgesic and Side Effects Concept in Lower Abdominal Surgical Oncology Procedures
Brief Title: Epidural Steroids With Intrathecal Nalbuphine for Lower Abdominal Oncologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R/17.04.127
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Lower Abdominal Oncologic Surgery

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-nalbuphine (Placebo Comparator): Epidural injection of normal saline followed with intrathecal injection of 0.6 mg nalbuphine in conjunction with 4 ml of hyperbaric bupivacaine 0.5%
  Interventions: Drug: Placebo-nalbuphine
- Dexamethasone-nalbuphine (Active Comparator): Epidural injection of dexamethasone followed with intrathecal injection of 0.6 mg nalbuphine in conjunction with 4 ml of hyperbaric bupivacaine 0.5%
  Interventions: Drug: Dexamethasone-nalbuphine

INTERVENTIONS:
Drug: Placebo-nalbuphine — Epidural injection of normal saline followed with intrathecal injection of 0.6 mg nalbuphine in conjunction with 4 ml of hyperbaric bupivacaine 0.5%
  Arms: Placebo-nalbuphine
Drug: Dexamethasone-nalbuphine — Epidural injection of dexamethasone followed with intrathecal injection of 0.6 mg nalbuphine in conjunction with 4 ml of hyperbaric bupivacaine 0.5%
  Arms: Dexamethasone-nalbuphine

SUMMARY:
Intraoperative pain, nausea, vomiting, hypotension, bradycardia are known side effects during lower abdominal surgery under spinal anesthesia, Time to 2 segment regression of sensory block and duration of effective analgesia prolonged with intrathecal (IT) 0.4 mg nalbuphine & IT 0.8 mg nalbuphine, but the incidence of side-effects was significantly higher with IT 0.8 mg nalbuphine compared with (IT) 0.4 mg nalbuphine.

DETAILED DESCRIPTION:
So, the hypothesis of using IT nalbuphine mid away dose 0.6 mg between the best intraoperative analgesic effective dose 0.8 mg and the least side effect producing dose 0.4mg with the addition of epidural dexamethasone could augment the postoperative analgesia and reduce the unwanted side effects. Epidural dexamethasone in a full dose of 8 mg is probably more effective than lower doses to control moderate to severe post-operative pain. Dexamethasone 8mg dose is surgically safe neither produced delayed wound healing nor elevated blood glucose level.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I or II.
* Undergoing laparotomy
* Undergoing oophorectomy
* Undergoing hysterectomy
* Undergoing rectal mass excision

Exclusion Criteria:

* Patient refusal.
* Hypersensitivity to amide local anesthetics.
* General contraindications to spinal anesthesia.
* Cardiac diseases.
* Hepatic failure.
* Renal failure.
* Respiratory failure.
* Communication barriers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-07 (Actual)

PRIMARY OUTCOMES:
Pain score | For 24 hours after surgery
  Pain visual analog score (0: no pain, 100: worst imaginable pain)

SECONDARY OUTCOMES:
Nausea and vomiting | For 24 hours after surgery
  (0: no nausea, 1: nausea, 2: mild vomiting, 3: moderate vomiting, 4: severe vomiting)
Sensory recovery | For 5 hours after induction of anaesthesia
  Regression to S1 spinal segment as tested with cold sensation
Motor recovery | For 5 hours after induction of anaesthesia
  The time until decreased a modified Bromage score of 0 (i.e. full leg movement)
First analgesic request | For 12 hours after induction of anaesthesia
  Time to first request of rescue analgesic
Intraoperative heart rate changes | For 3 hours after induction of anaesthesia
  Changes in heart rate during surgery
Intraoperative mean arterial blood pressure changes | For 3 hours after induction of anaesthesia
  Changes in mean arterial blood pressure during surgery
Postoperative heart rate changes | For 24 hours after surgery
  Changes in heart rate after surgery
Postoperative mean arterial blood pressure changes | For 24 hours after surgery
  Changes in mean arterial blood pressure after surgery
Cumulative use of antiemetic | for 24 hrs after surgery
  Cumulative use of metoclopramide and ondansetron after surgery
Cumulative use of rescue intravenous ketorolac | for 24 hrs after surgery
  Rescue use of ketorolac in case of severe pain conditions
Cumulative use of rescue intravenous nalbuphine | For 24 hours after surgery
  Rescue use of nalbuphine in case of severe pain conditions

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Ghanem, MD, Study Chair — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Faculty of Medicine, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided